CLINICAL TRIAL: NCT02212301
Title: Comparison of Two Marketed Lenses in a Controlled Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-5573
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Results first posted 2016-09-27 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-09

CONDITIONS: Eye Dryness
MeSH Terms: conditions — Xerophthalmia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- senofilcon A / lotrafilcon B (Active Comparator): Subjects were randomized to one of two lens wear sequences. Subjects randomized to this sequence first wore the senofilcon A contact lens and then wore the lotrafilcon B contact lens.
  Interventions: Device: senofilcon A; Device: lotrafilcon B
- lotrafilon B/ senofilcon A (Active Comparator): Subjects were randomized to one of two lens wear sequences. Subjects randomized to this sequence first wore the lotrafilcon B contact lens and then wore the senofilcon A contact lens
  Interventions: Device: senofilcon A; Device: lotrafilcon B

INTERVENTIONS:
Device: senofilcon A — Each study contact lens will be worn as daily wear modality for a period of 2 weeks each.
Device: lotrafilcon B — Each study contact lens will be worn as daily wear modality for a period of 2 weeks each.

SUMMARY:
This study is comparing two silicone hydrogel contact lenses in a controlled environment for identification of characteristics associated to vision.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be 18 years of age and less than 51 years of age;
2. The subject must have read and understood the Participant Information Sheet;
3. The subject must have read, signed and dated the Informed Consent;
4. The subject must be a current planned replacement soft contact lens wearer;
5. The subject must be a regular user of devices (computer, tablet and/or smart phone) for a minimum average of 5 ± 1 hours per day in a typical week
6. The subject must have a refractive error within the range of correction of both study contact lenses;
7. The subject must have a best-corrected visual acuity of 6/9 (20/30, 0.18 LogMAR) or better in each eye;
8. The subject must demonstrate an acceptable fit with both study contact lenses;
9. The subject must agree to wear their contact lenses as directed for the duration of the study (every day or for at least a minimum of five days per week for a minimum of six hours per day and be willing and able to adhere to the instructions set in the clinical protocol and maintain the appointment schedule;
10. The subject must have normal eyes with the exception of the need for visual correction.

Exclusion Criteria:

1. Any known sensitivity or intolerance to any of the contact lenses or adjunct products to be used.
2. Monocular vision (only one eye with functional vision or only one eye fitted with contact lenses).
3. Use of systemic or ocular concomitant medications which, as determined by the investigator, might contraindicate or interfere with contact lens wear.
4. Ocular anterior segment infection, inflammation, abnormality, or active disease, which would contraindicate contact lens wear.
5. Any moderate or severe ocular condition observed during slit lamp examination at the enrollment visit.
6. A history of herpetic keratitis, ocular surgery or irregular cornea(s).
7. Known pregnancy or lactation during the study period.
8. Enrollment of investigator's office staff, relatives, or members of their respective households.
9. Participation in any clinical trial within 30 days of the enrollment visit.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 45 subjects were enrolled into this study. Of the enrolled subjects 43 were dispensed and 2 subjects did not meet the eligibility criteria. Of the 43 dispensed subjects, 1 subject was discontinued 42 subjects completed the study.
Groups:
- Senofilcon A/ Lotrafilcon B: Subjects that received the senofilcon A contact lens in the first period and then received the lotrafilcon B contact lens in the second period.
- Lotrafilcon B / Senofilcon A: Subjects that received the lotrafilcon B contact lens in the first period and then received the senofilcon A contact lens in the second period.
Period: Period 1
Arm/Group | Senofilcon A/ Lotrafilcon B | Lotrafilcon B / Senofilcon A
Started | 21 | 22
Completed | 21 | 21
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Period 2
Arm/Group | Senofilcon A/ Lotrafilcon B | Lotrafilcon B / Senofilcon A
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed at least one study lens.
Groups:
- Dispensed Subjects: All subjects that were dispensed at least one lens throughout the duration of the study.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.1 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 14
Region of Enrollment [Number; unit: participants]
  United Kingdom | 43

OUTCOME MEASURES:

1. Primary Outcome: Tear Film Kinetics
Description: The non-invasive tear film break-up-time (NIBUT) is the time elapsed (in seconds) between eye opening after a blink, and the appearance of the first dark spot within the tear film when observed with the wide diffuse light source of the Tearscope. This measurement is indicative of the tear film stability and the on eye wettability of contact lenses.
Time Frame: 8 hour post insertion
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation (per-protocol). One subjects was excluded from the analysis population due to a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Senofilcon A: Subjects that received the senofilcon A contact lens in either the first or second period of the study.
- Lotrafilcon B: Subjects that received the lotrafilcon B in either the first or second period of the study.
Arm/Group | Senofilcon A | Lotrafilcon B
Number analyzed (Participants) | 41 | 41
Seconds | 5.590 (4.2705) | 6.941 (6.1257)

2. Primary Outcome: Time Controlled Visual Acuity
Description: The Time Controlled Visual Acuity test is a proprietary test part of MG Vision Advanced Visual Performance Assessment. The test for distance vision is carried out at 4m under high contrast and dim luminance. The test is presented on a fast response 17" LCD screen (1280 by 1064). The test for intermediate vision is carried out at 64cm under high contrast dim luminance. The test was presented on a fast response 13.3" LCD screen (3200 by 1800). Visual acuity will be measured in a controlled environment using logMAR units.
Time Frame: 8 hours post insertion
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation. The analysis was conducted for each lens at both near (40cm) and far distance (4m).
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Lotrafilcon B: Subjects that received the lotrafilcon B contact lens in either the first or second period of the study.
Arm/Group | Senofilcon A | Lotrafilcon B
Number analyzed (Participants) | 41 | 41
LogMAR
  Distance | -0.06 (0.092) | -0.07 (0.075)
  Intermediate | 0.07 (0.077) | 0.06 (0.074)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 1 month per subject.
Arm/Group | Senofilcon A | Lotrafilcon B
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 3/43 | 4/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Senofilcon A (N=43) | Lotrafilcon B (N=43)
Cold (General disorders) | 3 (3) | 4 (5) — Non-ocular adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less